CLINICAL TRIAL: NCT00157274
Title: Phase II Study of Alemtuzumab in Patients With Advanced Mycosis Fungoides/Sezary Syndrome
Brief Title: Study of Alemtuzumab to Treat Advanced Mycosis Fungoides/Sezary Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Latin American Cooperative Onco-Haematology Group - Peru (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MF/SS
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2007-04-03 (Estimated); Status verified 2005-09

CONDITIONS: Mycosis Fungoides; Sezary Syndrome
Keywords: Alemtuzumab; Mycosis fungoides; Sezary
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome | interventions — Alemtuzumab

INTERVENTIONS:
Drug: alemtuzumab

SUMMARY:
The investigators designed a compassionate basis phase II study for refractory/relapsed mycosis fungoides/Sezary syndrome consisting of alemtuzumab (Campath) for primary evaluation of overall response and time to relapse. Other goals to consider are toxicity and time to new therapy.

DETAILED DESCRIPTION:
* 20 relapsed or refractory advanced mycosis fungoides/Sezary syndrome patients are scheduled with gradually escalated doses (3 mg, 10 mg , and 30 mg) on sequential days during the first week, followed by 30 mg three times a week until 12 weeks.
* Patients must have serology negative for human T-lymphotropic virus 1 (HTLV-1) and until three different regimens of chemotherapy.
* Follow up for one year after last cycle of alemtuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Liver and renal function test less than twice upper label
* No active infection
* Written informed consent
* One to three regimens of previous chemotherapies

Exclusion Criteria:

* Abnormal renal or hepatic function
* Mycosis fungoides/Sezary syndrome in transformation
* HIV +
* HTLV-1 +
* Pregnancy
* Lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-07; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Overall response
Time to relapse
Event free survival

SECONDARY OUTCOMES:
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Brady E Beltran, MD, Principal Investigator — LACOGH - PERU
Locations (1):
- Schering Peruana S.A., Lima, Lima Province, Peru

REFERENCES:
- [Result] Lundin J, Hagberg H, Repp R, Cavallin-Stahl E, Freden S, Juliusson G, Rosenblad E, Tjonnfjord G, Wiklund T, Osterborg A. Phase 2 study of alemtuzumab (anti-CD52 monoclonal antibody) in patients with advanced mycosis fungoides/Sezary syndrome. Blood. 2003 Jun 1;101(11):4267-72. doi: 10.1182/blood-2002-09-2802. Epub 2003 Jan 23. PMID 12543862